CLINICAL TRIAL: NCT02467829
Title: What Are the Effects of Altering Handle Height of Posterior Walkers on Gait Parameters in Children With Spastic Cerebral Palsy?
Brief Title: Effects of Altering Handle Height of Posterior Walkers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Birmingham (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: RG_15-057
Record Dates: First submitted 2015-06-05; First posted 2015-06-10 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Cerebral Palsy
Keywords: Cerebral Palsy; Walking Aids
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 10° of elbow flexion (No Intervention): This handle height is the nearest position the walker can be set to to achieve 10° of elbow flexion. Elbow flexion is measured with the child standing in their walker using an electronic goniometer.
- 30° of elbow flexion (Experimental): Increase in handle height. This handle height is the nearest position the walker can be set to to achieve 30° of elbow flexion.
  Interventions: Device: Increase in handle height
- 50° of elbow flexion (Experimental): Increase in handle height. This handle height is the nearest position the walker can be set to to achieve 50° of elbow flexion.
  Interventions: Device: Increase in handle height

INTERVENTIONS:
Device: Increase in handle height — Elbow flexion is measured with the child standing in their walker using an electronic goniometer. Approximately 10° of elbow flexion is current recommended practice. 30° and 50° are increased handle heights.
  Arms: 30° of elbow flexion; 50° of elbow flexion

SUMMARY:
The aims of this study are to investigate what effect altering handle height of posterior walkers has on forces through the walker, posture, efficiency, stability, speed, turning and comfort, and to obtain data which helps therapists understand the bio-mechanics involved during use and if this alters depending on age, posture or strength. All participants will have cerebral palsy. This will allow informed prescription of walkers and identify potential for redesign to improve efficiency, promote strengthening or improve posture to maximise children's potential to continue functional walking into adulthood.

DETAILED DESCRIPTION:
Children with cerebral palsy (CP) find walking effortful due to weakness, lack of coordination between muscle groups, postural changes, poor balance and altered muscle tone. Walking aids improve efficiency, stability and posture.Posterior walkers were developed in the mid 1980's. There is evidence of their advantages over more traditional anterior walkers, however there is no evidence relating to setting handle height, and little information about bio-mechanics during use.

This is a quantitative pilot study with a cross over design. A purposive sample of approximately 15 children will be recruited from Birmingham Community Healthcare National Health Service (NHS) Trust. Assessments will be carried out at 3 different handle heights, determined by measuring elbow flexion when the participant is standing holding the handles of their walker. Participants will attend two assessments. One at their school, and a second at the University of Birmingham. Forces going through the walker and the participant's feet, range of motion at the trunk, hip and knee, velocity, step and stride length, double support time, physiological cost index, pain, gross motor function, hip abductor strength and ease of turning will be measured.

Analysis of variance with repeated measures will be used to analyse changes across handle heights and multiple linear regression to show associations between the dependent variables studied and identify potential confounding factors. p<0.05 will be considered statistically significant. Effect sizes needed for clinical significance will be considered.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of spastic Cerebral Palsy by a medical practitioner from clinical presentation.
* Aged 5-18 years.
* Able to walk 50m with a posterior walker without rest.
* Uses a posterior walker at least once a week.

Exclusion Criteria:

* Aged below 5 years or over 18.
* Orthopaedic surgery in the last 6 months, serial casting or botulinum toxin injections in the 12 weeks prior to or during the study, as gait could vary significantly following these interventions.
* Unable to walk 50m in a straight line and follow verbal prompts to turn.
* Insufficient understanding, in the opinion of their carer or therapist, to complete Faces rating scale.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-04 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Three dimensional gait analysis | Half a day
  Kinetic data will be captured using a 13 camera Vicon three dimensional motion analysis system. Reflective markers will be placed bilaterally on the acromion process, lateral epicondyle of the elbow, styloid process of the ulna, greater trochanter of the femur, anterior superior iliac spine, posterior superior iliac spine, lateral epicondyle of the femur, lateral malleolus, insertion of the achilles tendon and head of the fifth metatarsal. Markers will be placed on the corners of walker, at the top and bottom of it (8 in total). Trunk hip and knee angles on both sides of the body will be recorded throughout the gait cycle, as children with CP often have asymmetrical gait. Velocity, step and stride length and double support time will also be calculated using this system.

SECONDARY OUTCOMES:
Force through the legs of the walker and the participants feet. | Half a day
  A sensor will be placed in each of the four walker legs to measure the force going through each one. The force the participants's feet exert on the floor will be measured as they cross the force plate.
Physiological cost index | Half a day
  This measures efficiency of gait in beats per metre.It is calculated using the following formula:
  Walking heart rate-resting heart rate/walking speed. Heart rate is measured in beats/minute and speed in metres/minute. Heart rate will be continuously monitored electronically. It will be calculated over a distance of 50m.
The Faces Pain Scale -Revised | Half a day
  The participant chooses from one of 5 faces to indicate how much pain they are in. This will be repeated at each handle height.
Gross Motor function measure - 88 | 1-2 hours
  Used to assess change in gross motor function over time in children with CP. Participants are asked to do a series of simple tasks across 5 domains of lying and rolling, sitting, crawling and kneeling, standing, walking running and jumping.
Hip abductor strength | 10 mins
  Hip abductor strength will be measured in supine lying using a Kin Com dynamometer, as previously described by Engsberg at al (Engsberg et al., 2002).
Posterior walker 180 degree turn test | 5 mins
  This test has been designed for the purposes of this study. A line is taped on the floor perpendicular to the direction in which the participant is walking. They approach the line from a minimum of 3m away and turn when they reach the line. Direction of the turn (clockwise/anticlockwise), time and number of steps taken to turn 180 degrees is recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Marilyn Poole, BSc, Principal Investigator — Birmingham Community Healthcare NHS Trust
Locations (1):
- Kinesiology Laboratory, Birmingham, West Midlands, United Kingdom

REFERENCES:
- [Background] Greiner BM, Czerniecki JM, Deitz JC. Gait parameters of children with spastic diplegia: a comparison of effects of posterior and anterior walkers. Arch Phys Med Rehabil. 1993 Apr;74(4):381-5. PMID 8466419
- [Background] Logan L, Byers-Hinkley K, Ciccone CD. Anterior versus posterior walkers: a gait analysis study. Dev Med Child Neurol. 1990 Dec;32(12):1044-8. doi: 10.1111/j.1469-8749.1990.tb08521.x. PMID 2149558
- [Background] Mattsson E, Andersson C. Oxygen cost, walking speed, and perceived exertion in children with cerebral palsy when walking with anterior and posterior walkers. Dev Med Child Neurol. 1997 Oct;39(10):671-6. doi: 10.1111/j.1469-8749.1997.tb07361.x. PMID 9352728
- [Background] Park ES, Park CI, Kim JY. Comparison of anterior and posterior walkers with respect to gait parameters and energy expenditure of children with spastic diplegic cerebral palsy. Yonsei Med J. 2001 Apr;42(2):180-4. doi: 10.3349/ymj.2001.42.2.180. PMID 11371104
- [Background] Konop KA, Strifling KM, Wang M, Cao K, Schwab JP, Eastwood D, Jackson S, Ackman JD, Harris GF. A biomechanical analysis of upper extremity kinetics in children with cerebral palsy using anterior and posterior walkers. Gait Posture. 2009 Oct;30(3):364-9. doi: 10.1016/j.gaitpost.2009.06.012. Epub 2009 Jul 18. PMID 19616952
- [Background] Konop KA, Strifling KM, Wang M, Cao K, Eastwood D, Jackson S, Ackman J, Altiok H, Schwab J, Harris GF. [Upper extremity kinetics and energy expenditure during walker-assisted gait in children with cerebral palsy]. Acta Orthop Traumatol Turc. 2009 Mar-Apr;43(2):156-64. doi: 10.3944/AOTT.2009.156. Turkish. PMID 19448356
- [Background] Tomlinson D, von Baeyer CL, Stinson JN, Sung L. A systematic review of faces scales for the self-report of pain intensity in children. Pediatrics. 2010 Nov;126(5):e1168-98. doi: 10.1542/peds.2010-1609. Epub 2010 Oct 4. PMID 20921070
- [Background] Raja K, Joseph B, Benjamin S, Minocha V, Rana B. Physiological cost index in cerebral palsy: its role in evaluating the efficiency of ambulation. J Pediatr Orthop. 2007 Mar;27(2):130-6. doi: 10.1097/01.bpb.0000242440.96434.26. PMID 17314635
- [Background] Ketelaar M, Vermeer A, Helders PJ. Functional motor abilities of children with cerebral palsy: a systematic literature review of assessment measures. Clin Rehabil. 1998 Oct;12(5):369-80. doi: 10.1191/026921598673571117. PMID 9796927